CLINICAL TRIAL: NCT00144534
Title: An Open-label, Extension, Phase III Study to Evaluate the Long-term Safety and Efficacy of MRA in Patients With RA Who Participated in Study MRA213JP
Brief Title: Long-term Treatment Study of MRA for Rheumatoid Arthritis (RA) From Study MRA213JP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA215JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MRA (Tocilizumab)

INTERVENTIONS:
Drug: MRA (Tocilizumab) — 8mg/kg/4 weeks

SUMMARY:
This is an open-label, extension, Phase III study to evaluate the long-term safety and efficacy of MRA in patients with RA who participated in Study MRA213JP.

ELIGIBILITY:
Inclusion criteria

* Either MRA or placebo was administered at least 3 times in the preceding study, and there were confirmed to be no problems with respect to safety.
* In the case of Patients whose participation in the current study was judged to be inappropriate because of problems in the preceding study with respect to safety, these Patients must have been in the methotrexate dose group in the preceding study.

Exclusion criteria

* Administered drugs such as infliximab, etanercept, and leflunomide within 12 weeks before administration of the study drug
* Evaluated as belonging to Steinbrocker's class IV within 4 weeks before administration of the study drug
* Have not been registered by 3 months after the full code-breaking of the preceding study
* Were administered plasma exchange therapy between initiation of the preceding study and the initial administration in the current study
* Treated surgically (except for local surgery) within 4 weeks before administration of the study drug

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Efficacy:the frequency of amelioration of at least 20% in terms of the ACR criteria | throughout study
Frequency and degree (severity and seriousness) of adverse events and adverse drug reactions | throughout study
Pharmacokinetics of the serum MRA concentration | 0W,4W,8W,12W,LOBS

SECONDARY OUTCOMES:
Efficacy:time courses of DAS28, frequencies of amelioration of at least 20%, 50%, and 70% in terms of the ACR criteria, each item in the ACR core set | 0W,4W,8W,12W,LOBS

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical